CLINICAL TRIAL: NCT03402763
Title: Intervention to Promote Advance Care Planning for Older Adults in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-3371
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Emergency Medicine; Advance Care Planning
Keywords: Advance care planning; Older adults; Emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Participants will (1) be given either a short informational handout on the process and choices involved in advanced care planning or (2) be shown a less 6 minute video describing CPR, breathing tube placement and mechanical breathing support in addition to the general process of advanced care planning.
Masking Description: All patients and researchers are aware if the patient receives a handout or watches the ACP video.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Participants receive a short informational handout on the process and choices involved in advance care planning.
- Intervention (Experimental): Participants are shown a 6-minute video that describe CPR, breathing tube placement, and mechanical breathing support in addition to the general process of advance care planning.
  Interventions: Behavioral: Educational Video; Behavioral: Primary Care Provider Email

INTERVENTIONS:
Behavioral: Educational Video — The intervention is an educational video presented to patients in the ED with the intent to promote ACP among older adults.
  Arms: Intervention
Behavioral: Primary Care Provider Email — For intervention patients, an email will be sent to primary care providers explaining that the patient has seen a video about advance care planning, providing a synopsis of the video, and giving instructions about how to document end-of-life care preferences in the electronic health record.
  Arms: Intervention

SUMMARY:
There is an urgent need to increase advance care planning among older adults in order to ensure that patients receive care of the end of life that is consistent with their values and preferences. Emergency departments (EDs) provide an opportunity to reach a large proportion of older adults who have not yet completed advance care planning at a time when they are likely to recognize the need for such planning. The purpose of this pilot is to examine the potential of a video-supported intervention initiated during the emergency department visit to promote advance care planning.

DETAILED DESCRIPTION:
The overarching goal of this project is to understand the impact of an ED-initiated intervention on the promotion of advance care planning (ACP) among older adults. Participants are given either a short informational handout on the process and choices involved in ACP or watch a 6-minute video about ACP. The video describes cardiopulmonary resuscitation (CPR), breathing tube placement, and mechanical breathing support in addition to the general process of ACP. Following the video, patients in the intervention will also have an email sent to their primary care provider. The email will inform the primary care provider that the patient has watched a video about ACP, include a brief synopsis of the video, and provide instructions as to how to document the patient's preferences in the hospital's electronic health record in a way that will be accessible to other providers. Outcomes will include documentation of end-of-life care preferences in the electronic health records and patient-reported conversation with their provider as well as conversations with loved ones.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Ability to communicate in English
* Age 65-79 years with a serious medical illness: (1) Established diagnosis of metastatic cancer, advanced heart failure, chronic obstructive lung disease, end stage liver disease, end stage renal disease, (2) Unable to walk or requires human assistance with walking, (3) Two hospitalizations within the last 6 months
* Age 80 years or older

Exclusion Criteria:

* Critically ill (emergency severity index = 1)
* Cognitively impaired based on Six Item Screener < 4 or lack the capacity to consent
* Currently enrolled in hospice or comfort care program
* No working phone number
* Non English speaker

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Documentation of end-of-life preferences in the electronic health record | 3 months
  Since the ED visit, does the patient have any new preferences about CPR, intubation, or palliative care documented in their electronic health record?

SECONDARY OUTCOMES:
Conversation with Regular Provider | 3 months
  Patient-reported conversation with their regular provider (primary care physician, admitting physician, other outpatient provider) about what they would want done if they became very sick, had serious breathing trouble, heart stopped, or they could not make medical decisions from him or herself.
Conversation with Loved One | 3 months
  Patient-reported conversation with a trusted loved one (spouse, children, or sibling) about what they would want done if they became very sick, had serious breathing trouble, heart stopped, or they could not make medical decisions from him or herself.

OTHER OUTCOMES:
CPR and Intubation Preferences | 3 months
  Patient-reported preferences about if they would want CPR if heart stopped or intubation if patient could not breathe.
CPR Knowledge | 3 months
  True and false questions assessing patient knowledge about CPR.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F Platts-Mills, MD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: Yes
We plan to upload the data from the study on Open Science Framework.
Time Frame: Data will be uploaded within 1 year of study completion.